CLINICAL TRIAL: NCT00412100
Title: A Randomsied, Double-blind, Double-dummy, Parallel-group Multicentre Study to Demonstrate Improvement in Symptoms of Constipation in Subjects With Non-malignant Pain Taking Oxycodone Equivalent of 60-80 mg/Day as Oxycodone/Naloxone Prolonged Release Compared to Subjects Taking Oxycodone Prolonged Release Tablets Alone
Brief Title: Oxycodone-naloxone Prolonged Release Tablets in Relieving Opioid-related Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma Research GmbH & Co KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OXN3006; 2005-003510-15
Record Dates: First submitted 2006-12-14; First posted 2006-12-15 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Pain
Keywords: A randomised; double-blind; double-dummy; parallel-group multicentre study to demonstrate improvement in symptoms of constipation; Moderate to severe, chronic non-malignant pain
MeSH Terms: conditions — Pain

INTERVENTIONS:
Drug: Oxycodone naloxone prolonged release tablets (OXN)

SUMMARY:
The primary objective is to demonstrate that patients taking oxycodone/naloxone prolonged release tablets have improvement in symptoms of constipation compared to subjects taking oxycodone prolonged release tablets alone.

DETAILED DESCRIPTION:
Patients with a documented history of moderate to severe non-malignant pain that require around-the-clock opioid therapy will be randomised to an oxycodone or an oxycodone-naloxone treatment arm. The primary objective is to demonstrate that patients taking oxycodone/naloxone prolonged release tablets have improvement in symptoms of constipation compared to subjects taking oxycodone prolonged release tablets alone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects at least 18 years or older with moderate to severe pain that requires around the clock opioid therapy. Subjects must report constipation caused or aggravated by opioids.

Exclusion Criteria:

* Females who are pregnant or lactating.
* Subjects with evidence of any clinically unstable disease or subjects with evidence of impaired liver/kidney function upon entry into the study.
* Subjects with evidence of significant structural abnormalities of the gastrointestinal tract.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-04; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To demonstrate that subjects with moderate to severe non malignant pain taking oxycodone/naloxone prolonged release tablets have improvement in symptoms of constipation compared to subjects taking oxycodone prolonged release tablets alone. | 12 weeks with a 6 month open label extension

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Lowenstein, Principal Investigator — Private Practice

REFERENCES:
- [Derived] Lowenstein O, Leyendecker P, Lux EA, Blagden M, Simpson KH, Hopp M, Bosse B, Reimer K. Efficacy and safety of combined prolonged-release oxycodone and naloxone in the management of moderate/severe chronic non-malignant pain: results of a prospectively designed pooled analysis of two randomised, double-blind clinical trials. BMC Clin Pharmacol. 2010 Sep 29;10:12. doi: 10.1186/1472-6904-10-12. PMID 20920236
- See also: Results available on website — https://www.clinicaltrialsregister.eu/ctr-search/search?query=OXN3001